CLINICAL TRIAL: NCT02039817
Title: An Open-Label Pharmacokinetic and Pharmacodynamic Study of a Single Dose of IDN-6556 in Subjects With Severe Renal Impairment and in Matched Healthy Volunteers
Brief Title: PK and PD Study of IDN-6556 in Subjects With Severe Renal Impairment and Matched Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDN-6556-05
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-12

CONDITIONS: Renal Impairment; Renal Insufficiency; Kidney Disease; Kidney Diseases
Keywords: pharmacokinetics; pharmacodynamics; renal impairment
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Experimental): All subjects receive a single 50 mg oral dose of IDN-6556
  Interventions: Drug: IDN-6556
- Severe Renal Impairment (Experimental): All subjects receive a single 50 mg oral dose of IDN-6556
  Interventions: Drug: IDN-6556

INTERVENTIONS:
Drug: IDN-6556
  Other Names: emricasan; PF-03491390

SUMMARY:
This is an open-label, parallel-group study to compare the pharmacokinetics and pharmacodynamics of IDN-6556 following a single 50 mg oral dose of IDN-6556 in subjects with severe renal impairment and matched healthy volunteers with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Male or female subjects 18 - 75 years of age, able to provide written informed consent, understand and comply with all scheduled visits, and other requirements of the study
* Body mass index (BMI) 18.0 - 40.0 kg/m2 and body weight >50 kg
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from screening to one month after the last dose of study drug

Matched Healthy Volunteers:

* Medically healthy as determined by the Investigator
* Screening creatinine clearance ≥90 mL/min using the Cockcroft-Gault equation
* Supine blood pressure ≤145/90 mmHg
* No significant uncontrolled systemic or major illness that, in the opinion of the Investigator, would preclude the subject from participating in and completing the study
* Demographically comparable to subjects with severe renal impairment as follows:

  1. Mean body weight within ±10 kg
  2. Mean age within ±5 years
  3. Similar gender ratio

Severe Renal Impaired Subjects:

* Screening creatinine clearance (CLCR) <30 mL/min using the Cockcroft-Gault equation
* Supine blood pressure ≤170/110 mmHg
* Documented renal impairment indicated by reduced creatinine clearance within 12 months of screening or longer
* Stable renal function as evidenced by ≤30% difference in two measurements of creatinine clearance on two separate occasions separated by at least 28 days with one measurement being the value at screening.

Exclusion Criteria:

* History of renal trasplant
* Acute renal failure
* Subjects undergoing any method of dialysis or hemofiltration
* Evidence or history of clinically significant uncontrolled hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal product (e.g., inflammatory bowel disease, resections of the small or large intestine, etc.)
* History of febrile illness within 5 days prior to dosing
* Evidence of clinically significant liver disease or liver damage (e.g., hepatitis B or C, autoimmune hepatitis, primary biliary cirrhosis, non-alcoholic fatty liver disease, elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) that is considered clinically significant by the Investigator, etc.)
* Known infection with human immunodeficiency virus (HIV) upon serological testing
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QT or QTc interval of >480 milliseconds (msec) for subjects with severe renal impairment or >450 msec for matched healthy volunteers
* Subjects with active or history of malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Hagerty, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (2):
- United States (2):
  - Avail Clinical Research, DeLand, Florida
  - University of Miami, Miami, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, multicenter, parallel-group study to compare the PK and PD of IDN 6556 following a single 50 mg oral dose of IDN-6556 in subjects with severe renal impairment and matched subjects with normal renal function (healthy volunteers).
Pre-assignment Details: In total, 16 subjects were enrolled and dosed (8 subjects with severe renal impairment, and 8 healthy volunteers) with one 50mg dose of IDN-6556.
Groups:
- Healthy Volumteers: Healthy volunteers were given a single 50mg dose of IDN-6556
- Severe Renal Impairment: Severe Renal Impairment subjects were given a single 50mg dose of IDN-6556
Period: Overall Study
Arm/Group | Healthy Volumteers | Severe Renal Impairment
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Health Volunteers received one 50mg dose of IDN-6556
- Severe Renal Impairment: Severe Renal Impairment subjects received one 50mg dose of IDN-6556
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Median (Full Range); unit: years] | 61.0 [51 to 69] | 64.0 [54 to 68] | 62.0 [51 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: Area under the plasma concentration curve (AUC) parameters include AUC0-12, AUCinf, AUClast
Time Frame: 48 hours
Population: 7 subjects were used in the calculation of AUC0-inf for the healthy volunteer group as one subject had no identifiable terminal log-linear phase.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Healthy Volunteers; Severe Renal Impairment: Subjects received a single 50 mg oral dose of IDN-6556
Arm/Group | Healthy Volunteers | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8
h*ng/mL
  AUC 0-12 (h*ng/mL) | 102.0 (39.4) | 168.9 (42.3)
  AUC 0-inf (h*ng/mL) | 107.4 (41.3) | 188.5 (43.8)
  AUC last (h*ng/mL) | 105.9 (38.3) | 186.5 (43.4)

2. Secondary Outcome: Levels of cCK18
Description: Biomarker cCK18 (Cleaved cytokeratin 18) PK evaluations from pre-dose to 48 hours
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Healthy Volunteers | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8
U/L
  predose | 240.0 [165.5 to 336.0] | 223.5 [155.0 to 288.5]
  .5 hour | 201.5 [154.0 to 298.5] | 202.5 [178.5 to 300.0]
  1 hour | 208.0 [154.5 to 266.0] | 191.5 [183.0 to 283.0]
  2 hours | 202.5 [157.0 to 234.0] | 198.0 [175.5 to 284.0]
  3 hours | 184.5 [140.5 to 210.0] | 201.0 [190.5 to 295.0]
  4 hours | 183.5 [142.5 to 207.0] | 198.5 [178.5 to 284.5]
  5 hours | 179.0 [141.5 to 232.0] | 221.5 [162.0 to 291.5]
  8 hours | 178.0 [137.0 to 244.0] | 212.0 [152.5 to 256.5]
  12 hours | 167.0 [132.0 to 220.0] | 205.5 [155.0 to 266.0]
  24 hours | 204.0 [144.0 to 286.5] | 192.5 [159.5 to 266.0]
  48 hours | 206.5 [159.0 to 291.0] | 195.0 [183.0 to 295.0]

3. Primary Outcome: Cmax
Description: Maximum concentration (Cmax)
Time Frame: 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy Volunteers | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8
ng/mL | 28.5 (44) | 42.7 (57)

ADVERSE EVENTS:
Time Frame: 10 Days
Groups:
- IDN-6556: A single 50mg dose of IDN-6556
Arm/Group | IDN-6556
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less